CLINICAL TRIAL: NCT02212132
Title: Relations Between Cognitive Complaints and Cognitive Scores Goals in Cancer: Assessment of Metamemory
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: METACAN
Record Dates: First submitted 2014-08-04; First posted 2014-08-08 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Metamemory; Memory Complaints; Performance Mnemonic; Cancer
Keywords: metamemory; memory complaints; performance mnemonic; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient: Neuropsychological evaluation, psychopathological assessment and fatigue
  Interventions: Other: behavioral assessments
- Control group: Neuropsychological evaluation, psychopathological assessment and fatigue
  Interventions: Other: behavioral assessments

INTERVENTIONS:
Other: behavioral assessments — Neuropsychological evaluation, psychopathological assessment and fatigue

SUMMARY:
This pilot study is, in this new and original approach in cancer pathology, measure and explain the correspondence between perceived cognitive impairment (cognitive complaint) by cancer patients and their cognitive scores goals with tasks metamemory while controlling the anxiety and depression and fatigue factors of patients.

DETAILED DESCRIPTION:
The relationship between performance from neuropsychological tests and subjective complaints of cancer patients treated with chemotherapy or adjuvant hormone therapy is not clear, many studies have reported no significant correlation between these two measures: the perception of patients' their cognitive deficits is generally increased relative to that which is measured by neuropsychological testing.

The reason for this lack of association found is probably multifactorial. 1) It can be explained in part by methodological limitations in some studies (lack of sensitivity tests, experimental design). 2) psycho-order factors and fatigue are also an explanatory variable in the sense that literature data often show that cognitive complaints are correlated with levels of anxiety and depression and fatigue. 3) Finally, metacognition, often assessed in neurodegenerative diseases or even in normal aging to better understand its impact on cognitive disorders, including memory impairment, and the complaint has never been explored in patients with cancer.

Metacognition is a complex but highly sensitive to measure and understand the patient's complaint and correspondence or disagree with the actual performance concept. Metacognition refers A) metacognitive knowledge, ie knowledge of an individual's own cognitive processes; This is a non-dependent activity during which, upstream of the performance of any task, implement an appropriate strategy, anticipate and plan cognitive steps that would be necessary for its success general knowledge; and B) metacognitive experiences, ie knowledge that is based on a cognitive activity in progress, which allows to monitor and control the task in order to maintain or otherwise modify the cognitive processes involved.

While metacognitive knowledge (A) are assessed by multiple choice questionnaires, metacognitive experiences (B) allow targeted and precise fine measures of correspondence between the prediction performance by the patient himself and his actual performance a mnemonic task (for JOL and FOK Judgment of Learning for Feeling Of Knowing). Studies exploring the effects of age on metamemory usually show a deficit of these metacognitive experiences in normal aging compared to young subjects.

Collected at the time of learning, JOL is a prediction of future performance for information that have just been learned. More specifically, when learning words, the subject must judge its ability to further free recall for each item (quantitative data). This prediction is then compared to the actual memory performance found in the free recall task. This comparison allows to judge the accuracy of the prediction and therefore the accuracy of metamemory judgment.

The FOK corresponds to a prediction of performance information that could not be provided in free recall recognition. In practice, when an item is not recovered in free recall, the subject must judge its ability to recognize the correct answer among distractor responses.

Metacognitive processes can refer to the field of memory (metamemory) or attention (métaattention), but for now metamemory was much valued neuropsychological tests and the testing and are most successful and many more.

ELIGIBILITY:
Inclusion Criteria:

* Patient being treated for a solid or hematologic malignancy;
* Patients under 65 years of age;
* Patients Grade 3 'end primary school "minimum (scale Barbizet);
* Primary cancer of the central nervous system or brain metastases Absence;
* No major cognitive disorders;
* Lack of previous neurological;
* Lack of personality disorders and evolutionary psychiatric pathology.

Exclusion Criteria:

* Patients with paraneoplastic syndrome;
* Scalable psychiatric pathology;
* Refusal to participate;
* Patients unable to meet the cognitive tests;
* Use of drugs;
* Heavy drinking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient being treated for a solid tumor or hematological
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of metamemory through questionnaires | At study entry
  Comparison with questionnaires completed by healthy subjects matched controls.

SECONDARY OUTCOMES:
Influence of anxiety and depression and fatigue factors on metamemory. | At study entry
  Search by questionnaires the influence of anxiety and depression and fatigue factors on metamemory.

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, PhD, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François Baclesse, Caen, France